CLINICAL TRIAL: NCT06022497
Title: The Effect of Tidal Model-Based Emotion Regulation Nursing Interventions on Recovery in Individuals Diagnosed With Nursing Diagnosis of Impaired Mood Regulation
Brief Title: Tidal Model's Effects on Emotion Regulation and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gulsenay TAS SOYLU, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB Number: 21-11T/23
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Emotional Regulation; Psychiatric Nursing; Tidal Model; Recovery
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, Tidal Model-based emotion regulation nursing interventions were applied in addition to the routine treatment. Tidal Model-based emotion regulation nursing interventions were structured as eight sessions in total. Each individual in the intervention group participated in a session for a total of 8 weeks, one session per week. All interviews were conducted face to face.
  Interventions: Other: Tidal Model Based Emotion Regulation Interventions
- Control Group (No Intervention): The control group received only routine treatment.

INTERVENTIONS:
Other: Tidal Model Based Emotion Regulation Interventions — The Tidal Model is a nursing model and was developed by Phil Barker. It is an important model for psychiatric nursing care. In the research, nursing interventions for emotion regulation were structured by using the Tidal Model.At each session, emotion regulation interventions were applied within the Tidal Model care domains.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to investigate the effectiveness of Tidal Model-based emotion regulation interventions on recovery in individuals diagnosed with depression and nursing diagnosis of impaired mood regulation. The research was designed as a randomized controlled trial.

The main hypothesis; After nursing interventions for emotion regulation based on the Tidal Model, there is a significant difference between the recovery, difficulty in emotion regulation, depression levels and nursing outcome criteria of individuals in the intervention and control groups.

DETAILED DESCRIPTION:
The research carried out with patients followed in psychiatry outpatient clinics. As a result of the G-power analysis, the sample consisted of 23 interventions and 23 control groups. In the study, while the control group received only routine treatment, in the intervention group, Tidal Model-based nursing interventions were applied in addition to the routine treatment. Pre-tests administered before individuals were randomly assigned to the intervention and control groups. Randomization was created using the website randomizer.org. After this randomization was created, it was hidden from the physician who made the diagnosis of depression and from the researcher who conducted the interviews (allocation concealment). After the pre-tests were completed, the researcher (consulting faculty member) who knew the random assignment order was reached and the individuals were randomly assigned to the control or intervention group. Tidal Model-based nursing interventions were structured as 8 sessions in total. Each individual in the intervention group participated in a session for a total of 8 weeks, one session per week. In the eighth session, post-tests were applied to the individuals in the intervention group. Individuals in the control group were asked to come back 8 weeks after the first interviews and post-tests were applied. All interviews were conducted face to face. Recovery Assessment Scale (RAS), Difficulties in Emotion Regulation Scale (DERS), and Nursing Outcomes Criteria (NOC) were used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate Depression according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-V criteria
* Having a nursing diagnosis of Impaired Mood Regulation
* Psychiatrist prescribing serotonin reuptake inhibitor (SSRI)
* Man or Women aged 25-55
* Being followed by the psychiatry outpatient clinic
* Able to provide written informed consent

Exclusion Criteria:

* Presence of an additional mental illness
* Diagnosis of severe Depression according to DSM-V criteria
* Presence of suicidal attempts or thoughts
* Presence of another physical illness that affects cognition
* Have received any kind of therapy in the last six months
* Voluntary involvement in another study at the same time
* Inability to read and write

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Recovery Assesment Scale | before and end of the interventions (eight weeks)
  Recovery Assesment Scale was developed by Corrigan et al. (2004), and adapted to Turkish by Guler and Gurkan (2017) who also carried out the validity and reliability. It consist of 24 items, 5 point likert type. A high total score from the scale indicates a high level of improvement.Scale has five factors: personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, and no domination by symptoms
Difficulties in Emotion Regulation | before and end of the interventions (eight weeks)
  Difficulties in Emotion Regulation was developed by Gratz and Roemer (2004), and adapted to Turkish by Rugancı and Gencoz (2010) who also carried out the validity and reliability. It consist of 36 items, 5 point likert type. A high score on the scale indicates difficulty in emotion regulation. Scale has six factors: Awareness, Clarity, Impulse, Goals, Non-acceptance, Strategies.
Hamilton Depression Rating Scale | before and end of the interventions (eight weeks)
  Hamilton Depression Rating Scale was developed Hamilton et al. (1960), and adapted to Turkish by Akdemir et al. (1997) who also carried out the validity and reliability. The highest 51 points can be obtained from the scale.A score of less than 7 indicates that there is no depression, 8 to 15 points of mild depression, 16-28 points of moderate level, and 29 points and above indicate severe depression.

SECONDARY OUTCOMES:
Nursing Outcome Criteria | before and end of the interventions (eight weeks)
  Nursing Outcome Criteria is used to evaluate the patient's condition and is scored on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mahire Olcay Çam, Prof. Dr., Study Director — Ege University, Faculty of Nursing, Department of Pschiatric Nursing; Gulsenay TAS SOYLU, Principal Investigator — Izmir KAtip Celebi University, Faculty of Health Sciences, Department of Pschiatric Nursing
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Izmir, Bornova
  - Izmir Katip Celebi University, Izmir, Cigli

IPD SHARING:
Plan to Share IPD: No